CLINICAL TRIAL: NCT02225951
Title: A Randomised, Controlled, Open-label Trial to Investigate the Effect of a New Nutritional Supplement on Postprandial Glucose Response in Women Diagnosed With Gestational Diabetes Mellitus.
Brief Title: Meal Tolerance Trial in Pregnant Women Diagnosed With Gestational Diabetes Mellitus.
Acronym: GDM-MTT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Current protocol is not optimal/feasible
Sponsor: Danone Asia Pacific Holdings Pte, Ltd. (Industry)
Collaborators: Nutricia Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GDM.1.C/A
Record Dates: First submitted 2014-08-25; First posted 2014-08-26 (Estimated); Last update posted 2017-09-07 (Actual); Status verified 2017-09

CONDITIONS: Gestational Diabetes Mellitus in Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test group (Active Comparator): Nutritional product as breakfast.
  Interventions: Dietary Supplement: Nutritional product
- Control Group (Other): Standard breakfast according to ADA recommendations for pregnant women diagnosed with Gestational Diabetes Mellitus.
  Interventions: Other: Standard breakfast according to ADA recommendations

INTERVENTIONS:
Dietary Supplement: Nutritional product
  Arms: Test group
Other: Standard breakfast according to ADA recommendations
  Arms: Control Group

SUMMARY:
This study is initiated to investigate the effect of a nutritional product on the 3-hr postprandial glucose response compared to a control standard breakfast at baseline and after 4 weeks of intervention.

DETAILED DESCRIPTION:
The primary objective of the study is to investigate the effect of study product on the 3-hour postprandial glucose response compared to a controlled standard breakfast at baseline and after 4 weeks of intervention. Secondary objectives include investigation on the effect of the product compared to a control standard breakfast to the 3-hr postprandial insulin response, postprandial peak and delta peak concentration of glucose and insulin, fasting concentration of glucose and insulin, and insulin resistance as calculated by the HOMA index. The study also aims to measure compliance, study product intake and appreciation, safety and tolerance to study product, as well as satiety, daily energy and nutrient intake.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women, aged 18-40 years
2. 18.5 kg/m2 < pre-pregnancy BMI < 27.5 kg/m2 [representing low to moderate risk category, adapted from WHO expert panel recommendation on BMI categories for determining public health and clinical action (REF: Lancet, 2004)]
3. Singleton pregnancy
4. Newly GDM diagnosed women between 24 to (the latest) 32 weeks of gestation;
5. Diagnosed GDM according to either:

   * World Health Organization (WHO) criteria if one or more glucose values equal to or exceed these threshold values [75g Oral Glucose Tolerance Test: fasting 126 mg/dl; 2-h 140 mg/dl] or
   * American Diabetic Association (ADA) criteria if two or more glucose values equal to or exceed these threshold values [100g Oral Glucose Tolerance Test: fasting 95 mg/dl; 1-h 180 mg/dl; 2-h 155 mg/dl, 3-h 140/dl]
6. Willing and able to comply with the protocol
7. Signed informed consent

Exclusion Criteria:

1. Any gastrointestinal disease that interferes with bowel function and nutritional intake (i.e. constipation or diarrhea secondary to neuropathy, diarrhea due to chronic inflammatory bowel disease, gastroparesis, gastrectomy, galactosaemia, hyperemesis)
2. Currently on anti-diabetic therapy, for example on insulin or oral anti-diabetic medication
3. Already using a diabetes nutritional/dietary supplement (e.g. Glucerna®, Nutrient Diabetes®) within 4 weeks prior to signing informed consent
4. Known allergy or intolerance for any of the following ingredients; fish, milk, protein, lactose, fiber or soy
5. Any significant medical condition, other than GDM, that might interfere with the study or known to affect intra-uterine growth (e.g. Type 1 Diabetes, Type 2 Diabetes Mellitus, Crohn's disease, HIV/AIDS, liver disease, kidney disease etc.)
6. Currently or previously on special low/no carbohydrate diet (e.g. Atkin's diet) within 8 weeks prior to signing informed consent
7. Incapability to comply with study protocol or Investigator's uncertainty about the willingness or ability of the subject to comply with the protocol requirements
8. Participation in other studies involving investigational or marketed products concomitantly or within 4 weeks prior signing informed consent

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2014-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
3-hr postprandial glucose response | 28 days
  To investigate the effect of a nutritional product on the 3-hr postprandial glucose response compared to a control standard breakfast at baseline and after 4 weeks of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Kok Hian Tan, MBBS, Principal Investigator — KKH
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore